CLINICAL TRIAL: NCT04131673
Title: MS and NMOSD in African-Americans: a Prospective Data Collection Protocol Using REDCap
Brief Title: MS and NMOSD in African-Americans
Status: Withdrawn | Type: Observational
Why Stopped: IRB closed
Sponsor: Jagannadha R Avasarala (Other)
Responsible Party: Sponsor-Investigator, Jagannadha R Avasarala, Professor of Neurology, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 51232
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica
Keywords: multiple sclerosis; MS; Neuromyelitis optica spectrum disorder; NMOSD; African Americans
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African Americans with MS: African American patients seen in the University of Kentucky's Multiple Sclerosis Clinic between the ages of 18 and 80 who have been diagnosed with MS

SUMMARY:
This is a prospective study that aims to collect and review neuromyelitis optica spectrum disorder (NMOSD) data from African American patients with a known diagnosis of multiple sclerosis (MS). It is an investigational study, prospective in nature. No randomization of patients will be done. Information collected includes: Age, gender, age at diagnosis, MRI data (access to images), clinical presentation, findings on clinical examination, lab (blood and evoked potentials) and LP test results, eye exam findings if any and treatment, if started. Additional details may include other NEUROLOGICAL diseases which are also diagnosed (if any).

DETAILED DESCRIPTION:
African-Americans with MS are high risk for ambulatory difficulty given aggressive disease phenotype. Disease responsiveness to FDA-approved drugs is also marginal at best.

A positive correlation between the presence of oligoclonal bands (OCBs) and progressive course of MS has been established even when adjusted for ethnicity. It is well documented that the CSF humoral immune response, including a higher IgG index is higher in African-American MS patients. Although MRI lesions, specifically cord and infra-tentorial regions, contribute to disability, the phenotype in African-American populations is also probably linked to HLA-antigen complex. No study has ever collected data as it relates to ethnic background and MS. The University of Kentucky would be the first institution to collect such data.

This is a prospective study that will collect data from patients with the known diagnosis of MS who were later classified as NMOSD from the University of Kentucky's Multiple Sclerosis Clinic. Researchers will use REDCap to store data.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18 and 80
* are African-American
* have a diagnosis of MS and later diagnosis of NMOSD
* have been seen at the University of Kentucky's Kentucky Neuroscience Institute

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American patients who have been diagnosed with MS and later diagnosed as having NMOSD. They will be patients that have been seen in the Kentucky Neuroscience Institute (KNI). The age range will be 18-80.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical data collection and comparison | Through study completion, average duration of four years
  Collect patient age, sex, date of birth, and date of diagnosis to examine trends among this population.

SECONDARY OUTCOMES:
MRI analysis | Through study completion, average duration of four years
  Analyze MRIs of subjects to see how lesions contribute to this disorder over the course of the study.
Diagnostic tests collection and comparison | Through study completion, average duration of four years
  Collect blood tests, CSF studies, mimic conditions, and AQP4 testing will be collected and analyzed for changes over the course of the study and compared to other patients in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jagannadha Avasarala, MD PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No